CLINICAL TRIAL: NCT04737837
Title: A Multi-center,Open-label Real-world Study to Evaluate the Efficacy and Pharmaco-economics of Lacosamide as First Add-on Therapy for Adults and Children With Focal Onset Seizures
Brief Title: A Real World Study on the Efficacy and Safety of Lacosamide as Add-on Therapy for Focal-onset Epilepsy
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Jiangxi Qingfeng Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Other Study IDs: QF-LCM2020-1
Record Dates: First submitted 2021-01-24; First posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Epilepsy; Focal-Onset Seizure
Keywords: focal onset,lacosamide,CEA,Real-world,first add on
MeSH Terms: conditions — Epilepsy; Seizures | interventions — Lacosamide

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 26 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- children: Children aged 4~16 years with focal onset seizures
  Interventions: Drug: lacosamide
- Adult: Adults aged >16 years with focal onset seizures
  Interventions: Drug: lacosamide

INTERVENTIONS:
Drug: lacosamide — lacosamide as first add on therapy
  Other Names: Xinkang

SUMMARY:
The purpose of this trial is to evaluate the efficacy, safety, and pharmaco-economics of Lacosamide Tablet as first add-on therapy for uncontrolled focal onset epilepsy ,invetigating effects of lacosamide Tablet on cognitive function of children and anxiety and depression of adults with focal onset seizures In real-world clinical setting

DETAILED DESCRIPTION:
In many real world, lacosamide as the first add-on therapy can significantly improve the seizure freedom rate. Moreover, many pharmacoeconomic studies in Sweden and the United States have confirmed that lacosamide is a more cost-effective option.This is a real-world study to evaluate the efficacy, safety and cost-effectiveness of Generic lacoxamide tablets in the treatment of patients with focal epilepsy. During the trial, patients with focal epilepsy were treated with lacosamide for the first time after the failure of the original antiepileptic drug. At the same time, the cost-effectiveness of Generic lacosamide was evaluated from the perspective of economics, in order to provide the basis for the clinical choice for Chinese epilepsy patients.

ELIGIBILITY:
Inclusion Criteria:

* Before the start of the trial, to obtain the informed consent approved by the ethics committee voluntarily signed by each subject. For underage subjects, the informed consent jointly signed by the subjects themselves (≥10 years ) and their parents or legal guardian (in which the underage needs the signature with their parents or legal guardian, and the underage is defined as the subject under 18 years of age) ;
* Male and female, between the ages of 4 and 75 years;
* Diagnostic criteria of focal onset seizures (with or without focal to bilateral tonic clonic seizures) was based on the 2017 Classification of Epileptic Seizures from the International League Against Epilepsy (ILAE);
* In the 4 weeks before enrollment and during the baseline period, patients have been on only one stable dosage of antiepileptic drug and suitable for lacosamide add-on therapy according to their investigators criteria;
* During the 8-week retrospective baseline period, patients must have had at least 4 focal onset seizures per 28 days on average.

Exclusion Criteria:

* Patients had received previous lacosamide treatment;
* Female patients are pregnant, breast-feeding, and will not use contraception during the trial;
* Patients had known allergies to lacosamide or any ingredients of the drug, or with allergic constitution;
* Patients have a history of status epilepticus in the last 12 months;
* History of chronic alcohol or drug abuse; 6.history of suicide attempt or suicidal ideation in the past 6 months;
* Current use of Antidepressants, anxiolytics or antipsychotics;
* Patients suffer from progressive diseases that affect the patient's brain and its function;
* Sychogenic nonepileptic seizures;
* Patients suffer from serious lung and blood system diseases, malignant tumor, lower immune function and psychosis;
* Patients wil receive ketogenic diet therapy, or Four weeks before entering the screening period, patients used other drugs that may affect the absorption, distribution, metabolism and excretion of lacosamide, such as antipsychotics, monoamine oxidase inhibitors, barbiturates (except for combined use as anticonvulsant therapy), narcotic analgesics.
* Patients Had epilepsy brain surgery, or will undergo epilepsy surgery in the next four months.
* Investigators considered Patients as unsuitable for this trial.

Ages: 4 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Adult and children patients (aged 4~75 years) with uncontrolled focal onset seizures and receiving only one baseline AED
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-31 (Estimated); Primary Completion 2021-11-28 (Estimated); Study Completion 2022-02-28 (Estimated)

PRIMARY OUTCOMES:
The change in seizure frequency per 4 week from retrospective baseline to the maintenance period | up to 26 weeks
  The seizure frequency is standardized to a 4 week duration
≥50responder rate | up to 26 weeks
  percentage of subjects with a 50 % or greater reduction in seizure frequency per 4 weeks from retrospective baseline to maintenance

SECONDARY OUTCOMES:
Seizure freedom rate | up to 26 weeks
  percentage of subjects who achieved seizure-free during maintenance period
Retention rate | up to 26 weeks
  the percentage of patients continuing lacosamide at the end of a specified period
Cognitive function | up to 26 weeks
  Cognitive function in elderly children aged greater than or equal to 6 years is assessed by Wechsler Intelligence Scale for Children-Revised (WISC-RC) ;
Cognitive function | up to 26 weeks
  Cognitive function in young children aged less than 6 years is assessed by Chinese Wechsler Young Children scale of Intelligence(C - WYCSI)
Evaluation for anxiety status | up to 24 weeks
  using by seven-item Generalized Anxiety Disorder scale (GAD-7)
Evaluation for depression status | up to 24 weeks
  using by Neurological Disorders Depression Inventory for Epilepsy(NDDI-E)

OTHER OUTCOMES:
the Cost of epilepsy treatment | up to 26 weeks
  To calculate the direct medical costs, including personal expenses and medical insurance reimbursement expenses, mainly include examination expenses, disposal expenses, medicine expenses, hospitalization expenses and other expenses
Cost-Effectiveness Analysis(CEA） | up to 26 weeks
  CEA=cost/efficacy(C/E)

CONTACTS AND LOCATIONS:
Overall Officials: Dong Zhou, Doctor, Principal Investigator — West China Hospital
Locations (19):
- China (19):
  - Beijing Children's Hospital affiliated to Capital Medical University, Beijing, Beijing Municipality
  - The First Affiliated Hospital of Jinan University, Guangzhou, Guangdong
  - The Second Affiliated Hospital of Guangzhou Medical University, Guangzhou, Guangdong
  - Shenzhen Children's Hospital, Shenzhen, Guangdong
  - The First Affiliated Hospital of Zhengzhou University, Zhengzhou, Henan
  - Wuhan Union Hospital, Wuhan, Hubei
  - Xiangya Hospital of Central South University, Changsha, Hunan
  - Nanjing Brain Hospital, Nanjing, Jiangshu
  - The Children's Hospital Affiliated to Suzhou University, Suzhou, Jiangshu
  - Wuhan Children's Hospital, Wuhan, JiangShu
  - The First Hospital of Jilin University, Changchun, Jilin
  - The First Affiliated Hospital of China Medical University, Shenyang, Liaoning
  - Shandong Provincial Hospital, Jinan, Shandong
  - Huashan hospital affiliated to Fudan University, Shanghai, Shanghai Municipality
  - The Children's Hospital of Fudan University, Shanghai, Shanghai Municipality
  - The Second Affiliated Hospital of Xi'an Jiaotong University College of Medicine, Xi’an, Shanxi
  - West China Hospital of Sichuan University, Chengdu, Sichuan
  - West China Second Hospital of Sichuan University, Chengdu, Sichuan
  - Children's Hospital Affiliated to Medical College of Zhejiang University, Hangzhou, Zhejiang

IPD SHARING:
Plan to Share IPD: Undecided